CLINICAL TRIAL: NCT02966288
Title: A Randomized Controlled Trial to Assess the Pain-control Efficacy of Intra-articular Toradol Compared to Oral NSAIDs: A Pilot Study
Brief Title: A Trial to Assess the Pain-control Efficacy of Intra-articular Toradol Compared to Oral NSAIDs
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Kimberly A Chambers, Clinical Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0616
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Arthritic Knee Pain
MeSH Terms: interventions — Ketorolac Tromethamine; Ketorolac; Anti-Inflammatory Agents, Non-Steroidal; Ibuprofen

ARMS (2):
- Toradol injection (Experimental): 3-ml solution that contains 2 ml of normal saline and 1 ml of Toradol, 30 mg, will be infused into the affected joint.
  Interventions: Drug: Toradol
- Oral NSAID (Active Comparator): 800mg Motrin will be administered. (non-steroidal anti-inflammatory drug (NSAID))
  Interventions: Drug: Oral NSAID

INTERVENTIONS:
Drug: Toradol — 3-ml solution that contains 2 ml of normal saline and 1 ml of Toradol, 30 mg, will be infused into the affected joint.
  Other Names: ketorolac
  Arms: Toradol injection
Drug: Oral NSAID — 800mg Motrin will be administered. (non-steroidal anti-inflammatory drug (NSAID))
  Other Names: ibuprofen
  Arms: Oral NSAID

SUMMARY:
The study objective is to determine whether a single intra-articular dose of an anti-inflammatory (Toradol) will reduce the need for other analgesic medications and, if so, how long the benefits will last.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiographic evidence of osteoarthritis (OA) who present to the ED with a chief complaint of knee pain that the treating provider attributes to their arthritis.

Exclusion Criteria:

* Acute knee trauma
* Intra-articular steroid injection within 6 months
* History of gout or rheumatoid arthritis
* X ray evidence of pathologic fracture, malignancy, or other non-OA cause of symptoms
* Signs or symptoms or high risk of acute infection: Recent fevers and chills; Erythema, warmth, or pain out of proportion to exam; History of hemodialysis; History of IV drug use
* Lidocaine allergy
* Any contraindication to NSAID therapy, including: Allergy; Pregnancy; History of renal insufficiency; History of gastritis, GERD or GI bleeding; Primary care physician's restriction of its use
* Contraindication to the procedure, including: Hemophilia; History of total knee replacement of the affected joint
* An inability to give informed consent; Active psychosis; Diminished capacity requiring another person to provide consent for medical treatment
* An inability to be contacted for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Pain Medication Usage for Breakthrough Pain | 72 hours
Pain Level as Assessed by a Visual Analogue Scale | 72 hours

SECONDARY OUTCOMES:
Pain Medication Usage for Breakthrough Pain | 1 week post treatment
  The number of pills will be reported
Pain Medication Usage for Breakthrough Pain | 2 weeks post treatment
  The number of pills will be reported
Pain Medication Usage for Breakthrough Pain | 3 weeks post treatment
  The number of pills will be reported
Pain Medication Usage for Breakthrough Pain | 4 weeks post treatment
  The number of pills will be reported
Pain Level as Assessed by a Visual Analogue Scale | 1 week post treatment
Pain Level as Assessed by a Visual Analogue Scale | 2 weeks post treatment
Pain Level as Assessed by a Visual Analogue Scale | 3 weeks post treatment
Pain Level as Assessed by a Visual Analogue Scale | 4 weeks post treatment
Number of Participants who had a second visit to a Emergency Department or Clinic | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Chambers, MD, Principal Investigator — The University of Texas Health Science Center, Houston